CLINICAL TRIAL: NCT03746899
Title: Expanded Access to Provide Intramuscular Injections of PLX-PAD for the Treatment of Subjects With Critical Limb Ischemia (CLI) With Minor Tissue Loss Who Are Unsuitable for Revascularization
Brief Title: Expanded Access for Treatment Use of PLX-PAD in Critical Limb Ischemia (CLI)
Status: Available | Type: Expanded Access
Sponsor: WideTrial, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PLX-CLI-06
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Critical Limb Ischemia (CLI)
Keywords: Critical Limb Ischemia (CLI)
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: PLX-PAD — PLX-PAD cell therapy to be administered via 30 IM injections (0.5 mL each) to the index leg leg per treatment, in each of two treatments, 8 weeks apart

SUMMARY:
This is an Expanded Access program (EAP), sponsored by WideTrial for the treatment of critical limb ischemia (CLI).

Widetrial, an Expanded Access specialist, has arranged to supply participating sites with PLX-PAD for CLI patients who cannot participate in the ongoing research trial and who seek exploratory treatment options. This program includes FDA-authorized cost recovery, meaning payment is required to cover a portion of the costs of delivering product and complying with regulatory obligations.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female subjects between ages 45 to 99 years of age at the time of screening.
2. Subjects with a diagnosis of PAD due to atherosclerosis at the stage of CLI, with minor tissue loss up to the ankle level (ulcer/s and/or necrosis).
3. Ankle pressure (AP) ≤70 mmHg or toe pressure (TP) ≤50 mmHg in the index leg or transcutaneous oxygen pressure (TcPO2) ≤30 mmHg.
4. Subject unsuitable for revascularization (by any method) in the index leg based on unfavorable risk-benefit assessment of the physician investigator. Unsuitability to revascularization should be based on any of the following:

   1. Anatomic considerations as: inappropriate target artery, diffuse/extensive tibial and/or peroneal artery lesions, inadequate distal run-off.
   2. Technical considerations as: inappropriate bypass conduit, failed recent revascularization.
   3. Medical considerations: subject's comorbidities.
5. Signed informed consent form.
6. Subjects are not eligible for the ongoing phase III study with PLX-PAD in CLI (PLX-CLI-03) due to at least one of the following criteria:

   1. Evidence of active localized osteomyelitis secondary to contiguous focus of infection, unless amputation is expected within 1 month post PLX-PAD administration. In case of osteomyelitis, patients must be treated with antibiotics during screening and PLX-PAD administration or as long as there is evidence of active infection.
   2. Subject on renal replacement therapy or with eGFR <15 mL/min.
   3. Current treatment with high dose systemic steroids (prednisone equivalent >7.5 mg/day) or topical steroids on the index leg.
   4. History of autologous bone marrow transplantation (if not due to hematologic malignancy) or solid organ transplantation, clinically stable.
   5. Immunocompromised subjects due to disease for any reason, including immunosuppressive therapy, at screening (for steroid therapy, refer to the criterion c)
   6. CLI with major tissue loss (Rutherford Category 6) in the contralateral leg.
   7. Diabetes mellitus with glycosylated hemoglobin (HbA1c) >10% at Screening.
   8. HIV controlled by antiretroviral therapy
   9. Past drug or alcohol abuse. Known history of cancer is eligible if occurred beyond 2 years before screening

Exclusion Criteria:

1. Non-atherosclerotic PAD and vasculitis (e.g., Buerger's disease [thromboangiitis obliterans], Takayasu's arteritis, etc.).
2. CLI with major tissue loss (Rutherford Category 6) in the index leg. Ulcers from venous or neuropathic origin if not associated with at least one ulcer from arterial origin.
3. Evidence of active infection in either leg (e.g., cellulitis, myositis) except localized osteomyelitis secondary to contiguous focus of infection, under antibiotic treatment.
4. Subject having undergone surgical/endovascular revascularization or major/minor amputation, in either leg, less than 1 month prior to Screening.
5. Planned or potential need for major/minor amputation or any revascularization of either leg within 1 month of EAP entry upon physician's judgment.
6. Aortoiliac stenosis or common femoral artery stenosis ≥70%, or otherwise suspicion of inadequate inflow to the index leg at the time of Screening.
7. Current evidence or sign supporting an assessment of life expectancy of less than 6 months.
8. Stroke or acute myocardial infarction within 3 months prior to Screening.
9. Severe congestive heart failure symptoms (New York Heart Association [NYHA] Stage IV) at screening.
10. Life-threatening ventricular arrhythmia - except in subjects with an implantable cardiac defibrillator at screening.
11. Uncontrolled severe hypertension during Screening.
12. Current or history of proliferative retinopathy.
13. Known active Hepatitis B virus or Hepatitis C virus infections at Screening.
14. Acquired immunodeficiency syndrome (AIDS), severe uncontrolled inflammatory disease, or severe uncontrolled autoimmune disease (e.g., ulcerative colitis, Crohn's disease, etc.).
15. Subjects at an increased risk of blood clotting or bleeding according to the Physician's judgment.
16. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3×ULN. Subjects with higher levels may be included if the condition associated with the increase in those liver enzymes is known and is considered clinically stable.
17. Current drug or alcohol abuse.
18. Subject is currently enrolled in, or has not yet completed a period of at least 30 days since ending another investigational device or drug trial(s) unless in long-term follow-up phase (in which there is no IP administration).
19. Current use or use within 30 days prior to screening of wound dressing containing cells or growth factors like Apligraf®, or topical platelet derived growth factor.
20. Current use, planned use, or use within 15 days prior to treatment of hyperbaric oxygen therapy, spinal cord stimulation, or lumbar sympathectomy.
21. Exposure to allogeneic cell based therapy in the past or exposure to autologous cell therapy in the last 12 months before screening.
22. Known allergies to any of the following: dimethyl sulfoxide (DMSO), human serum albumin, bovine serum albumin.
23. History of allergic/hypersensitivity reaction to any substance having required hospitalization and/or treatment with intravenous steroids/epinephrine, known allergy to more than 3 allergens, or in the opinion of the Physician the subject is at high risk of developing severe allergic/hypersensitivity reactions.
24. History of severe atopic disease (including but not limited to chronic urticaria, respiratory allergy requiring oral steroids), or history of uncontrolled Asthma (Global Initiative for Asthma [GINA] III-IV).

    1. Pulmonary disease requiring supplemental oxygen treatment on a daily basis.
    2. History of acute transfusion reaction.
    3. History of allogeneic bone marrow transplantation.
    4. Active malignancy except for successfully resected skin basal cell carcinoma or not located on the index leg.
    5. Pregnant or lactation women
    6. Inability to understand and provide an informed consent.

Ages: 45 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult